CLINICAL TRIAL: NCT02884505
Title: Improving the Assessment of Hypersomnolence
Status: Completed | Type: Observational
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Other Study IDs: 2015-1462
Record Dates: First submitted 2016-08-16; First posted 2016-08-31 (Estimated); Last update posted 2019-08-22 (Actual); Status verified 2019-08

CONDITIONS: Disorders of Excessive Somnolence
MeSH Terms: conditions — Disorders of Excessive Somnolence | interventions — Evoked Potentials, Auditory

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with Hypersomnolence: Patients referred for polysomnography and multiple sleep latency test
  Interventions: Device: Pupillometry; Behavioral: Psychomotor Vigilance Task; Other: Auditory Evoked Potential; Behavioral: Hypersomnia Severity Index

INTERVENTIONS:
Device: Pupillometry — Measures pupillary dynamics in darkness and light conditions
Behavioral: Psychomotor Vigilance Task — Response time task measuring neurobehavioral alertness
Other: Auditory Evoked Potential — Measure of electroencephalographic response to standardized auditory tones
Behavioral: Hypersomnia Severity Index — Self-report measure of hypersomnolence

SUMMARY:
The overall purpose of this study is to employ a pragmatic, multidimensional assessment of hypersomnolence that "piggybacks" on routine clinical care in patients with suspected disorders of central nervous system (CNS) hypersomnia, to determine whether these additional objective and subjective assessments are useful in the diagnosis and management of these patients.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-89
* Referred for polysomnography/multiple sleep latency test at Wisconsin Sleep, the sleep medicine clinic and laboratory of the University of Wisconsin-Madison

Exclusion Criteria:

* unstable medical condition that, in the opinion of the investigators, would make it unsafe for the subject to participate

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients referred for polysomnography and multiple sleep latency test at the University of Wisconsin-Madison
Sampling Method: Non-Probability Sample
Enrollment: 132 (Actual)
Dates: Start 2017-08-25 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Proportion of Patients Categorized with Hypersomnolence | 2 Years
  Multiple measurements will be aggregated to arrive at the primary outcome of proportion of patients categorized as having hypersomnolence using either standard assessments or standard assessments plus additional novel hypersomnolence measures of pupillometry, psychomotor vigilance task, and auditory evoked potentials. Proportion of patients with hypersomnolence using standard measures will be calculated as number of patients with mean sleep latency (MSL) on multiple sleep latency test (MSLT) <8 minutes divided by total number of patients. Proportion of patients categorized as having hypersomnolence with additional novel hypersomnolence measures will be calculated as the number of patients with MSL<8 minutes, and/or pupillary unrest index (PUI) >8.9 on pupillometry, and/or PVT lapses >3, and/or P300 delay/sleep negativity during auditory evoked potentials divided by total number of patients.

CONTACTS AND LOCATIONS:
Overall Officials: David T Plante, MD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin-Madison, Department of Psychiatry, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No